CLINICAL TRIAL: NCT05909722
Title: Prospective, Multicentre Study to Validate the GastroIntestinal Dysfunction Score (GIDS) and Describe Prevalence, Outcomes, and Management of Phosphate Disorders in Intensive Care Patients
Brief Title: Validation of the GIDS and Description of Phosphate Disorders
Acronym: GUTPHOS
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Annika Reintam Blaser, Associate Professor, University of Tartu
Other Study IDs: GUTPHOS study
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Organ Dysfunction Scores; Hypophosphatemia
MeSH Terms: conditions — Hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gastrointestinal Dysfunction Score will be calculated — We collect routine daily data on GI signs and symptoms and calculate the score (GIDS). We collect serum phosphate values as measured in routine practice of participating sites.
  Other Names: Phosphate levels

SUMMARY:
This study will address two specific research questions simultaneously:

1. validation of the GastroIntestinal (GI) Dysfunction score (GIDS).
2. description of epidemiology, risk factors, and management of phosphate disorders.

The aim is to recruit 20 ICUs and 1500 ICU patients. Sites will recruit all consecutive adult patients to a maximum of 120 patients or a maximum recruitment period of 8 weeks, whichever comes first. Daily data collection on gastrointestinal signs and symptoms as well as phosphate values and management will be collected during ICU stay for maximum of 7 days. 28 and 90 day mortality and days free of organ support will be the main outcomes. Secondary outcomes include prevalence of hypo- and hyperphosphatemia and description of their management.

DETAILED DESCRIPTION:
Patient population All consecutive adult patients that are admitted to participating ICU during a recruitment period of maximum 8 weeks.

Duration of the study for the individual patient:

1. Study period of a maximum of 7 days
2. Follow-up period of a maximum of 90 days All patients will be included in the Part A of the study validating GIDS, patients from sites with routine serum phosphate measurements will be included also in the Part B of the study where additional data on serum phosphate levels and management of phosphate disorders will be collected. There will be no additional measurements due to study participation, daily routine is documented.

Baseline characteristics will be collected at ICU admission/study inclusion Daily data include routine data on organ dysfunctions and organ support therapies and specific data on phosphate where available.

Outcome data include 28 and 90 days mortality, and days free of organ support by day 28.

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU during the study period
* Age ≥18 years

Exclusion Criteria:

* Age <18 years;
* Patients with restrictions of care such as "no intubation" or "no renal replacement therapy" on ICU admission and patients admitted for treatment as organ donors;
* Continuous chronic home ventilation for neuromuscular disease;
* Declined participation or informed consent (if the local ethics committee requests the latter for this non-interventional study);
* Readmission to ICU during the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients that are admitted to participating ICU during a recruitment period of maximum 8 weeks. In all included patients data on organ dysfunctions will be collected, in patients from sites with routine serum phosphate measurements additional data on phosphate values and management will be collected (inclusion in the Phosphate part of the study).
Sampling Method: Probability Sample
Enrollment: 2681 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
90 days mortality | 90 days
  Survival status at 90 days after ICU admission
28 days mortality | 28 days
  Survival status at 28 days after ICU admission

SECONDARY OUTCOMES:
Days free of organ support | 28 days
  Days alive and free of organ support (including parenteral nutrition-free days) by day 28
Prevalence of phosphate disorders at ICU admission | Day of ICU admission (day 1)
  Prevalence of hypo- and hyperphosphatemia on ICU admission
Incidence of phosphate disorders during seven days of ICU stay | 7 days
  Incidence of hypo- and hyperphosphatemia during seven days of ICU stay
The amount of phosphate administered | 7 days
  The amount of phosphate administered to patients with hypophosphatemia
Change in serum phosphate level in response to phosphate supplementation | 7 days
  Chenge in serum phosphate level in response to phosphate supplementation (correction/overcorrection/no correction)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur van Zanten, PhD, Principal Investigator — Gelderse Valley Hospital
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reintam Blaser A, Padar M, Mandul M, Elke G, Engel C, Fischer K, Giabicani M, Gold T, Hess B, Hiesmayr M, Jakob SM, Loudet CI, Meesters DM, Mongkolpun W, Paugam-Burtz C, Poeze M, Preiser JC, Renberg M, Rooijackers O, Tamme K, Wernerman J, Starkopf J. Development of the Gastrointestinal Dysfunction Score (GIDS) for critically ill patients - A prospective multicenter observational study (iSOFA study). Clin Nutr. 2021 Aug;40(8):4932-4940. doi: 10.1016/j.clnu.2021.07.015. Epub 2021 Jul 18. PMID 34358839
- [Derived] Melchers M, Kouw IWK, Arabi YM, Casaer MP, Cotoia A, Gunst J, Malbrain MLNG, Schaller SJ, Starkopf J, Rehal MS, Blaser AR, van Zanten ARH. Prospective multicenter study to describe the prevalence, outcomes, and management of phosphate disorders in intensive care patients: Study protocol for part B of the international GUTPHOS study. Clin Nutr ESPEN. 2024 Oct;63:681-687. doi: 10.1016/j.clnesp.2024.07.024. Epub 2024 Jul 26. PMID 39069259
- [Derived] Kouw IWK, Melchers M, Mandul M, Arabi YM, Casaer MP, Cotoia A, Gunst J, Malbrain MLNG, Schaller SJ, Starkopf J, Sundstrom Rehal M, Reintam Blaser A, van Zanten ARH. Prospective multicenter study to validate the gastrointestinal dysfunction score (GIDS) in intensive care patients: Study protocol for Part A of the international GUTPHOS study. Clin Nutr ESPEN. 2024 Oct;63:702-708. doi: 10.1016/j.clnesp.2024.07.023. Epub 2024 Jul 26. PMID 39069258